CLINICAL TRIAL: NCT05723614
Title: TRUE HAVEN: TRUsted rEsidents and Housing Assistance to Decrease Violence Exposure in New Haven
Brief Title: TRUsted rEsidents and Housing Assistance to Decrease Violence Exposure in New Haven
Acronym: TRUE HAVEN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: 2000032184; 1R01MD017526-01 (NIH)
Record Dates: First submitted 2023-02-01; First posted 2023-02-13 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Firearm Injury
Keywords: gun violence; structural racism
MeSH Terms: conditions — Systemic Racism

STUDY DESIGN:
Intervention Model Description: One component of the intervention will focus on providing housing support for recently incarcerated people as well as family members of currently incarcerated people. The target sample size is about 1,400. The other component of the intervention is mental wellness training for neighborhood residents to participate in trauma-informed care training sessions.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention)
- Intervention (Experimental): The two components in the intervention arm of TRUE HAVEN are: housing support for recently incarcerated people as well as family members of currently incarcerated people, and mental wellness training for neighborhood residents to participate in trauma-informed care training sessions.
  Interventions: Behavioral: TRUE HAVEN

INTERVENTIONS:
Behavioral: TRUE HAVEN — The two components of the TRUE HAVEN intervention are: housing support for recently incarcerated people as well as family members of currently incarcerated people, and mental wellness training for neighborhood residents to participate in trauma-informed care training sessions.
  Arms: Intervention

SUMMARY:
The overall objective of this study is to implement and test a strengths-based, community-driven intervention to reduce gun violence by (1) improving housing stability through providing financial assistance coupled with comprehensive financial education for the re-entry population as well as their family members, and (2) fostering greater support for mental health by training a trusted network of community members in trauma-informed counseling.

DETAILED DESCRIPTION:
Proposed is a type I hybrid effectiveness/implementation study using a neighborhood-level, stepped-wedge trial design across six primarily Black/Latinx, socially vulnerable neighborhoods in New Haven. Residents of each neighborhood who have been affected by incarceration (i.e., currently have a family member incarcerated or a person returning to the community from prison within the last 12 months) will be eligible for our intervention for a period of 6 months. The Consolidated Framework for Implementation Research (CFIR) and the Reach, Effectiveness, Adoption, Implementation, and Maintenance (RE-AIM) implementation science frameworks will be used to measure and track processes in achieving outcomes. A mixed methods approach will be used, primarily the use of quantitative methods for this study, along with qualitative focus groups will be conducted to assess some implementation outcomes. The primary outcome, rates of gun violence at the neighborhood level, are obtained from administrative data. Survey data will be collected for some implementation process measures (e.g., assessing acceptability and appropriateness of the intervention).

ELIGIBILITY:
All residents in the study neighborhoods are eligible for outcome assessment. For the intervention component of housing support, the below inclusion and exclusion criteria apply.

Inclusion criteria:

* Age 18 or above
* Family member currently incarcerated or person returning from prison within the last 12 months
* Live in one of the six neighborhoods with highest rates of gun violence in New Haven, Connecticut

Exclusion criteria:

* Plans to leave the study area within 1 year

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 61770 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Change in rates of gun violence | Baseline, 6 months, 12 months, 18 months, 24 months, 30 months, and 36 months
  The neighborhood rate of incident gun violence assessed among everyone in the neighborhoods; these data will be provided annually by the New Haven Police Department.

SECONDARY OUTCOMES:
Change in neighborhood social cohesion using the Social Cohesion sub-scale of the Sampson Collective Efficacy Scale | Baseline, 6 months, 12 months, and 24 months
  This is a neighborhood-level outcome on residents' perception of the strengths of relationships and solidarity among their neighbors. Data will be provided annually from DataHaven based on a representative sample of approximately 1% of population across each neighborhood of New Haven. The measure is based on Social Cohesion sub-scale of the Sampson Collective Efficacy Scale, which is a 5-point scale (score range: 1(strongly disagree) to 5(strongly agree)).
Change in participant self-efficacy based on the Generalized Self-Efficacy Scale | Baseline, 6 months, 12 months, and 24 months
  Individual-level perceptions and reactions to life's situations will be measured using a survey among the about 1,400 recruited participants. The measure is based on the Generalized Self-Efficacy Scale, which is a 4-point scale (score range: 1(not at all true) to 4(exactly true)).
Change in perceived health and well-being based on the Well-being Assessment | Baseline, 6 months, 12 months, and 24 months
  Individual-level perceived health and well-being including dimensions of subjective well-being, general health, health problems, sense of direction and purpose in life, emotional support, and sense of belonging to community will be measured using a survey among the about 1,400 recruited participants. This composite measure is based on Well-being Assessment (Adult - 12 items) - 100 Million Healthier Lives. Each item is an 11-point scale (score range: 0(worst) to 10(best)). Higher scores indicate better perceived health and well-being.
Change in financial security | Baseline, 6 months, 12 months, and 24 months
  Financial readiness for an emergency will be assessed using a survey among the recruited participants. The measure is based on one 5-point item (score range: 1(worst) to 5(best)) measuring financial capability.

CONTACTS AND LOCATIONS:
Overall Officials: Emily Wang, MD, MAS, Principal Investigator — Yale University
Locations (4):
- United States (4):
  - Beaver Hills, New Haven, Connecticut
  - Fair Haven, New Haven, Connecticut
  - Hill North and South, New Haven, Connecticut
  - Newhallville, New Haven, Connecticut

IPD SHARING:
Plan to Share IPD: Yes
Deidentified data will be made publicly available following study completion.
Time Frame: One year following the end of the funding.
Access Criteria: One year after the end of study funding, the de-identified data will be available upon request to the principal investigators of the study (Brita Roy, Brita.Roy@nyulangone.org; Virginia Spell, vtspell@ulsc.org; Emily Wang, emily.wang@yale.edu)

REFERENCES:
- [Derived] Tong G, Spell VT, Horton N, Thornhill T, Keene D, Montgomery C, Spiegelman D, Wang EA, Roy B. Trusted residents and housing assistance to decrease violence exposure in New Haven (TRUE HAVEN): a strengths-based and community-driven stepped-wedge intervention to reduce gun violence. BMC Public Health. 2023 Aug 14;23(1):1545. doi: 10.1186/s12889-023-15997-x. PMID 37580653
- [Derived] Tong G, Spell VT, Horton N, Thornhill T, Keene D, Montgomery C, Spiegelman D, Wang EA, Roy B. TRUsted rEsidents and Housing Assistance to decrease Violence Exposure in New Haven (TRUE HAVEN): A strengths-based and community-driven stepped-wedge intervention to reduce gun violence. Res Sq [Preprint]. 2023 May 10:rs.3.rs-2874381. doi: 10.21203/rs.3.rs-2874381/v1. PMID 37214890